CLINICAL TRIAL: NCT01274260
Title: Steroids in Pediatric Acute Lung Injury/ARDS Trial: A Blinded, Placebo-controlled, Randomized Clinical Trial
Brief Title: Trial of Steroids in Pediatric Acute Lung Injury/ARDS
Acronym: SPALIT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Tennessee (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Steroids in Pediatic ALI/ARDS
Record Dates: First submitted 2011-01-09; First posted 2011-01-11 (Estimated); Last update posted 2014-05-28 (Estimated); Status verified 2014-05

CONDITIONS: Acute Respiratory Distress Syndrome (ARDS); Acute Lung Injury (ALI)
Keywords: child; infant; lung injury; inflammation; pneumonia; ventilator
MeSH Terms: conditions — Respiratory Distress Syndrome; Acute Lung Injury; Lung Injury; Inflammation; Pneumonia | interventions — Methylprednisolone; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental Group (Active Comparator): Intervention: Subjects in this study group will receive a loading dose of methylprednisolone 2mg/kg followed by 1mg/kg/day of methylprednisolone infusion from day 1 to day 7; 0.5mg/kg/d from days 8 to 10, 0.25mg/kg/d on days 11 and 12, 0.125mg/kg/d on days 13 and 14. The study drug infusion will be discontinued after 14 days.
  Interventions: Drug: methylprednisolone
- Placebo Group (Placebo Comparator): Intervention: The placebo will be 0.9% (normal) saline and the active medication will be diluted in 0.9% (normal) saline. The placebo group with receive the masked study drug in infusion rates that mimic the infusions received by the experimental group.
  Interventions: Drug: Normal Saline (0.9%)

INTERVENTIONS:
Drug: methylprednisolone — Subjects in this group will receive a loading dose of methylprednisolone 2mg/kg followed by 1mg/kg/day of methylprednisolone infusion from day 1 to day 7; 0.5mg/kg/d from days 8 to 10, 0.25mg/kg/d on days 11 and 12, 0.125mg/kg/d on days 13 and 14. The study drug infusion will be discontinued after 14 days.
  Arms: Experimental Group
Drug: Normal Saline (0.9%) — The placebo will be 0.9% (normal) saline and the active medication will be diluted in 0.9% (normal) saline.
  Arms: Placebo Group

SUMMARY:
Acute lung injury (ALI) and acute respiratory distress syndrome (ARDS) are devastating disorders associated with lung inflammation, low oxygen levels and respiratory failure in children. Prevalence of ALI ranges from 2.2 to 12 per 100,000 children per year. Using these estimates, up to 9,000 children each year will develop ALI/ARDS, which may cause upto 2,000 deaths per year. Currently, there are no specific therapies directed against ARDS/ALI in children. In adult patients, use of steroids early in the course of ARDS appears promising. There are no published clinical trials examining the use of steroids for the treatment of ALI/ARDS in children.

Hypothesis:

Subjects with ALI/ARDS receiving steroids early in the course of disease (within 72 hours) and longer than 7 days will have improved clinical outcomes as compared to placebo control group as defined by (a) a decreased duration of mechanical ventilation and (b) significantly increased PaO2/FiO2 ratios.

ELIGIBILITY:
Inclusion Criteria:

1. Between 1 month and 18 years of age; AND
2. Admitted to the PICU with a diagnosis of ALI or ARDS, as defined by:

   1. acute onset of the disease,
   2. PaO2/FiO2 ratio <300,
   3. evidence of bilateral infiltrates on chest radiography, and
   4. no evidence of cardiac dysfunction; AND
3. Intubated and mechanically ventilated.

Exclusion Criteria:

1. Underlying disease requiring steroids >0.5mg/kg/day of methylprednisolone (eg. Asthma)
2. HIV positive, or have any other congenital or acquired immunodeficiency;
3. Terminally ill patients or patients on hospice care or if there is a lack of commitment to aggressive intensive care
4. Cytotoxic therapy within the past 3 weeks
5. Major gastrointestinal bleeding within last 1 month
6. Extensive burns (>20% total body surface area of full- or partial-thickness burns)
7. Known or suspected adrenal insufficiency
8. Vasculitis or diffuse alveolar hemorrhage
9. Bone marrow or lung transplant
10. Disseminated fungal infections
11. Severe chronic liver disease
12. Other conditions with estimated 6-month mortality of 50% or higher

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2010-10; Primary Completion 2014-01 (Actual); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Duration of mechanical ventilation | 0-28 days
  Number of hours required for positive pressure ventilation after the start of study drug

SECONDARY OUTCOMES:
Improvement in oxygenation | 0-28 days
  Differences in the PaO2/FiO2 ratios between the two randomized groups
Incidence of nosocomial infections | 0-35 days
  Infection surveillance will be in the form of tracheal aspirate for gram stain and culture done prior to study entry and then every 3-5 days. If a subject spikes a fever during the study drug infusion, they will have blood, urine and tracheal aspirate cultures done along with CBC and CRP. Number of nosocomial infections documented via surveillance cultures will be compared between groups.
Incidence of hyperglycemia | 0-28 days
  Number of times that the subject has a Blood Glucose >180 mg/dL (10 mmol/L) will be compared between the randomized groups

CONTACTS AND LOCATIONS:
Locations (1):
- Le Bonheur Children's Hospital, Memphis, Tennessee, United States

REFERENCES:
- [Derived] Kimura D, Saravia J, Rovnaghi CR, Meduri GU, Schwingshackl A, Cormier SA, Anand KJ. Plasma Biomarker Analysis in Pediatric ARDS: Generating Future Framework from a Pilot Randomized Control Trial of Methylprednisolone: A Framework for Identifying Plasma Biomarkers Related to Clinical Outcomes in Pediatric ARDS. Front Pediatr. 2016 Mar 31;4:31. doi: 10.3389/fped.2016.00031. eCollection 2016. PMID 27066464
- [Derived] Schwingshackl A, Kimura D, Rovnaghi CR, Saravia JS, Cormier SA, Teng B, West AN, Meduri UG, Anand KJ. Regulation of inflammatory biomarkers by intravenous methylprednisolone in pediatric ARDS patients: Results from a double-blind, placebo-controlled randomized pilot trial. Cytokine. 2016 Jan;77:63-71. doi: 10.1016/j.cyto.2015.10.007. Epub 2015 Nov 3. PMID 26545141
- [Derived] Drago BB, Kimura D, Rovnaghi CR, Schwingshackl A, Rayburn M, Meduri GU, Anand KJ. Double-blind, placebo-controlled pilot randomized trial of methylprednisolone infusion in pediatric acute respiratory distress syndrome. Pediatr Crit Care Med. 2015 Mar;16(3):e74-81. doi: 10.1097/PCC.0000000000000349. PMID 25634565